CLINICAL TRIAL: NCT06149689
Title: mFOLFIRINOX Plus Radiotherapy to Patients With CA19-9-normal Advanced Pancreatic Cancer
Acronym: PTCA199-7
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-7
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mFOLFIRINOX plus radiotherapy (Experimental): Patients with advanced pancreatic adenocarcinoma will receive a modified FOLFIRINOX regimen (oxaliplatin [70 mg per square meter of body surface area], irinotecan [130 mg per square meter], leucovorin [200 mg per square meter], and fluorouracil [2000 mg per square meter] every 2 weeks). Four-week chemotherapy is considered as a cycle. Patients will be recommended to receive Intensity-Modulated Radiation Therapy (IMRT) after about 4~6 cycles of chemotherapy. The following treatment after radiotherapy will be applied according to the newest edition of National Comprehensive Cancer Network (NCCN) guideline.
  Interventions: Combination Product: mFOLFIRINOX plus radiotherapy

INTERVENTIONS:
Combination Product: mFOLFIRINOX plus radiotherapy — Patients with advanced pancreatic adenocarcinoma will receive a modified FOLFIRINOX regimen (oxaliplatin [70 mg per square meter of body surface area], irinotecan [130 mg per square meter], leucovorin [200 mg per square meter], and fluorouracil [2000 mg per square meter] every 2 weeks). Four-week chemotherapy is considered as a cycle. Patients will be recommended to receive Intensity-Modulated Radiation Therapy (IMRT) after about 4~6 cycles of chemotherapy. The following treatment after radiotherapy will be applied according to the newest edition of National Comprehensive Cancer Network (NCCN) guideline.
  Other Names: mFOLFIRINOX plus IMRT

SUMMARY:
The purpose of this study is to evaluate the efficacy of mFOLFIRINOX plus radiotherapy to Patients with CA19-9-normal Advanced Pancreatic Cancer.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. In 2011, the PRODIGE trial has shown that oxaliplatin, irinotecan, fluorouracil, and leucovorin (FOLFIRINOX) was associated with a survival advantage but had increased toxicity.

Carbohydrate antigen 19-9 (CA19-9) is the most widely used biomarker in pancreatic cancer. Circulating CA19-9 levels are positively correlated with tumor burden and stage in pancreatic cancer with a diagnostic sensitivity of approximately 80%, suggesting that approximately 20% of patients have normal CA19-9 levels. It is well recognized that Lewis (-) individuals, constituting approximately 10% of the population, have low or no secretion of CA19-9 due to the lack of critical enzyme involved in CA19-9 biosynthesis. Thus, approximately 10% of patients with pancreatic cancer have normal CA19-9 levels regardless of tumor stage. Our previously retrospective study has shown that CA19-9-normal advanced pancreatic cancer may be more sensitive to chemotherapy combined with radiotherapy.

The purpose of this study is to evaluate the efficacy of mFOLFIRINOX plus radiotherapy to patients with CA19-9-normal advanced pancreatic cancer. Progression-free survival (PFS), objective response rate (ORR), overall survival (OS) and disease control rate (DCR) are measured every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed advanced pancreas adenocarcinoma.
* Patients who have not received any form of anti-tumor therapy.
* Baseline serum CA19-9 ≤ 37 U/mL, CEA≤ 5.2 ng/mL, and CA125 ≤ 35 U/mL.
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* The expected survival ≥ 3 months.
* Adequate organ performance based on laboratory blood tests.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Pregnant or nursing women.
* Patients who have received any form of anti-tumor therapy.
* Baseline serum CA19-9 > 37 U/mL, CEA > 5.2 ng/mL, or CA125 > 35 U/mL.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
* Renal insufficiency or dialysis
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
* Patients who are allergic to oxaplatin or other chemotherapy drugs.
* Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival，OS | At the end of Cycle 1 (each cycle is 21 days)
  OS of subjects from recruiting to the time of death from any cause

SECONDARY OUTCOMES:
progression-free survival, PFS | At the end of Cycle 1 (each cycle is 21 days)
  PFS of subjects from recruiting to the time of disease progression
objective response rate (ORR) | At the end of Cycle 1 (each cycle is 21 days)
  CR + PR
disease control rate (DCR) | At the end of Cycle 1 (each cycle is 21 days)
  CR + PR + SD

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luo G, Liu C, Guo M, Long J, Liu Z, Xiao Z, Jin K, Cheng H, Lu Y, Ni Q, Yu X. CA19-9-Low&Lewis (+) pancreatic cancer: A unique subtype. Cancer Lett. 2017 Jan 28;385:46-50. doi: 10.1016/j.canlet.2016.10.046. Epub 2016 Nov 10. PMID 27840089
- [Background] Luo G, Jin K, Guo M, Cheng H, Liu Z, Xiao Z, Lu Y, Long J, Liu L, Xu J, Liu C, Gao Y, Ni Q, Yu X. Patients with normal-range CA19-9 levels represent a distinct subgroup of pancreatic cancer patients. Oncol Lett. 2017 Feb;13(2):881-886. doi: 10.3892/ol.2016.5501. Epub 2016 Dec 14. PMID 28356973
- [Background] Luo G, Liu C, Guo M, Cheng H, Lu Y, Jin K, Liu L, Long J, Xu J, Lu R, Ni Q, Yu X. Potential Biomarkers in Lewis Negative Patients With Pancreatic Cancer. Ann Surg. 2017 Apr;265(4):800-805. doi: 10.1097/SLA.0000000000001741. PMID 28267695